CLINICAL TRIAL: NCT04024930
Title: Endoscopic Ultrasound Guided Choledocoduodenostomy With the Lumen Apposing Metal Stent [Axios® Stent]
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI18_0034
Record Dates: First submitted 2019-07-12; First posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: EUS Guided Biliary Drainage
Keywords: EUS guided biliairy drainage; EUS Choledoco-duodenostomy; Axios stent; Lumen Apposing Metal Stent

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endoscopic Ultrasound (EUS) guided biliary drainage is indicated in case of impossibility or failure of classic biliary drainage by endoscopic retrograde cholangio-pancreatography (ERCP). Recently the investigators reported a good efficiency of EUS guided choledocoduodenostomy using the HOT-AXIOS device (Electrocautery enhanced lumen apposing metal stent) in a retrospective multicentric study. Utilization of the recommended technique (direct punction with the HOT AXIOS using a pure cut current + using a 6 mm Stent) was the only predicting factor of clinical success. The investigators reevaluate this procedure one year after in the same centers.

ELIGIBILITY:
Inclusion Criteria:

* patients with tumoral obstruction of the distal biliary tract that have been treated by an EUS-CDS with a electrocautery enhanced LAMS

Exclusion Criteria:

* < 18 years old
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with tumoral obstruction of the distal biliary tract that have been treated by an EUS-CDS with a electrocautery enhanced LAMS
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
technical success rate | Day 1
  Technical success was defined as the ability to correctly deploy the Hot AXIOS stent between the common bile duct and the duodenal bulb with visualization of bile flow

SECONDARY OUTCOMES:
Clinical success | Day 28
  Number of participants with a decrease in the bilirubin level ≥ 50% at day 7, or normalization at day 28
Periprocedural adverse events: adverse events that occur during the procedure | Day 1
  Number of participants with an adverse event occuring during the procedure of EUS-CDS. ASGE lexicon will be used to grade these adverse events.
short-term adverse events | Day 7
  Number of participants with an adverse event occuring between the procedure and discharge from hospital. Adverse events were rated according to the American Society for Gastrointestinal Endoscopy (ASGE) lexicon will be used to grade these adverse events.
Long-term biliary adverse events: biliary adverse events that occur after discharge from hospital. | Year 1
  Number of participants with a biliary adverse event occuring after discharge from hospital. Adverse events were rated according to the American Society for Gastrointestinal Endoscopy (ASGE) lexicon will be used to grade these adverse events.
Six month stent patency rate | Month 6
  rate of permeability of the stent 6 months after the procedure

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Hospital University, Brest
  - University Hospital, Limoges
  - Hospital Private Jean MERMOZ, Lyon
  - APHM Hospital La Timone, Marseille
  - University Hospital, Montpellier
  - APHP Hospital Saint-Antoine, Paris
  - Hospital Cournouaille, Quimper
  - Hospital Jacques Lacarin, Vichy